CLINICAL TRIAL: NCT02522000
Title: Symptom Perception in Patients With Functional Dyspepsia: Involvement of the TRPV-1 Neuropeptide Pathway
Brief Title: Functional Dyspepsia and Symptom Perception
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: METC142070
Record Dates: First submitted 2015-07-29; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-07

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with functional dyspepsia
- Healthy controls

SUMMARY:
Functional dyspepsia (FD) is a heterogeneous disorder with multifactorial pathophysiology. Patients with FD have visceral hypersensitivity to mechanical and chemical stimuli. Several previous studies have described an increased chemosensitivity to oral capsaicin ingestion. Capsaicin is a natural agonist of TRPV-1 receptors present on afferent sensory neurons. Activation of the TRPV-1 receptor by capsaicin or other agonists results in the release of several neuropeptides (i.e. substance P, somatostatin). Besides, increased duodenal permeability and disruption of tight junction structure in FD patients compared to healthy volunteers has been reported in a recent study. In this observational study investigators will evaluate the role of the TRPV-1 neuropeptide pathway in patients with functional dyspepsia and healthy controls.

ELIGIBILITY:
Healthy volunteers

Inclusion criteria:

- No gastrointestinal symptoms or history of gastrointestinal disease meeting ROME III criteria for functional dyspepsia and Irritable Bowel Syndrome (IBS).

Exclusion criteria:

* Inability to stop the intake of nonsteroidal antiinflammatory drugs (NSAIDs) within 14 days prior to endoscopy and within two days prior to multi-sugar test.
* Inability to stop the intake of medication affecting gastrointestinal function (e.g. proton pump inhibitors, prokinetics, laxatives) within 5 days prior to endoscopy, multi-sugar test and combined meal- and gastric emptying test
* Current use of antidepressants
* Medical history of diabetes mellitus
* Medical history of coeliac disease
* Organic disease at upper gastrointestinal endoscopy (i.e. erosive esophagitis, Barrett's esophagus, benign esophageal stricture, Schatzki ring, esophageal carcinoma, esophageal candidiasis, gastric ulcer, gastric erosions, gastric cancer, duodenal erosions or duodenal ulcer)
* First-degree family members with diabetes mellitus type I, coeliac disease, Crohn's disease or ulcerative colitis
* Medical history of food allergy or anamnestic evidence of food allergy
* Presence of coagulation disorders or use of the following anticoagulants: coumarin derivates, new oral anticoagulants (NOACs: dabigatran, apixaban and rivaroxaban), and clopidogrel (Patients or healthy controls using calcium carbasalate (acetylsalicylic acid 100mg 1dd1) are eligible to participate in the study. Patients or healthy controls using higher doses of calcium carbasalate will be excluded from the study).
* Dieting
* Pregnancy or lactation
* Smoking
* Excessive alcohol use (>20 alcoholic consumptions/week) and inability to avoid use of alcohol in the 2 days prior to endoscopy and multi-sugar test

Functional dyspepsia patients

Inclusion criteria:

- Patients referred for upper gastrointestinal endoscopy by either general practitioners or physicians from the gastroenterology outpatient clinic and meeting ROME III criteria for functional dyspepsia.

Exclusion criteria:

* Inability to stop the intake of nonsteroidal antiinflammatory drugs (NSAIDs) within 14 days prior to endoscopy and within two days prior to multi-sugar test.
* Inability to stop the intake of medication affecting gastrointestinal function (e.g. proton pump inhibitors, prokinetics, laxatives) within 5 days prior to endoscopy, multi-sugar test and combined meal- and gastric emptying test
* Current use of antidepressants
* Medical history of diabetes mellitus
* Medical history of coeliac disease
* Organic disease at upper gastrointestinal endoscopy (i.e. erosive esophagitis, Barrett's esophagus, benign esophageal stricture, Schatzki ring, esophageal carcinoma, esophageal candidiasis, gastric ulcer, gastric erosions, gastric cancer, duodenal erosions or duodenal ulcer)
* First-degree family members with diabetes mellitus type I, coeliac disease, Crohn's disease or ulcerative colitis
* Medical history of food allergy or anamnestic evidence of food allergy
* Presence of coagulation disorders or use of the following anticoagulants: coumarin derivates, new oral anticoagulants (NOACs: dabigatran, apixaban and rivaroxaban), and clopidogrel (Patients or healthy controls using calcium carbasalate (acetylsalicylic acid 100mg 1dd1) are eligible to participate in the study. Patients or healthy controls using higher doses of calcium carbasalate will be excluded from the study).
* Dieting
* Pregnancy or lactation
* Smoking
* Excessive alcohol use (>20 alcoholic consumptions/week) and inability to avoid use of alcohol in the 2 days prior to endoscopy and multi-sugar test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 patients with functional dyspepsia and 20 healthy controls will be included
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
TRPV-1 neuropeptide pathway (TRPV-1 and mucosal neuropeptides) | Test day 1: mucosal biopsies are taken during upper gastrointestinal endoscopy
  The primary outcome measure is the TRPV-1 neuropeptide pathway which includes both TRPV-1 and mucosal neuropeptide concentrations (e.g. substance P, somatostatin), assessed with real time polymerase chain reaction (PCR) and radioimmunoassay respectively.

SECONDARY OUTCOMES:
Symptom scores for psychopathology | 14-day period between testday 1 and testday 2
  The Patient Health Questionnaire 9 (PHQ-9) and GAD-7 questionnaires will be used for the assessment of depressive and anxiety disorders respectively.
  During 7 consecutive days a digital device will be carried out for assessment of symptoms several times a day (experience sampling method/ESM).
Symptom scores for dyspepsia | 14-day period between testday 1 and testday 2
  Dyspeptic symptoms will be measured with two questionnaires to acquire more detailed information about complaints in patients with functional dyspepsia. The dyspepsia symptom questionnaire and the symptom checklist of the Nepean Dyspepsia Index will be used to grade the presence and intensity of dyspeptic symptoms.
  In addition, participants will report dyspeptic symptoms during 14 consecutive days in an end-of-day diary.
  During 7 consecutive days a digital device will be carried out for assessment of symptoms several times a day (experience sampling method/ESM).
Symptom scores for quality of life | This questionnaire is fulfilled once, in the 14-day period between testday 1 and testday 2
  Quality of life will be assessed with the Health Survey 26 (SF-36) questionnaire.
Postprandial symptoms after ingestion of a standardized meal | Testday 2: Postprandial symptoms are scored using a Likert scale at 15-minute intervals for a period of 240 minutes postprandial.
In vivo gastroduodenal and small intestinal permeability | Day before testday 2
  Gastroduodenal en small intestinal permeability will be assessed with a multisugar test.
Transcription of genes encoding for proteins involved in mucosal barrier function and symptom perception | Testday 1: gastric and duodenal biopsies are taken during upper gastrointestinal endoscopy.
Serotonin metabolism in mucosal tissue | Testday 1: gastric and duodenal biopsies are taken during upper gastrointestinal endoscopy
Serotonin metabolism in plasm | Testday 2: blood samples for serotonin analyses are taken preprandial and every 30 minutes after intake of a standardized meal during 240 minutes postprandial.
Gastric emptying for solids using the 13C-sodium octanoate stable isotope breath test | Testday 2: Repeated measure: breath samples for analysis of gastric emptying are taken preprandial and every 15 minutes after intake of a standardized meal during 240 minutes postprandial.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Conchillo, MD, PhD, Principal Investigator — Maastricht University Medical Center, Maastricht, The Netherlands
Locations (3):
- Netherlands (3):
  - Maastricht University Medical Center (MUMC+), Maastricht
  - Zuyderland Medical Center, Sittard-Geleen
  - St. Elisabeth Medical Center, Tilburg